CLINICAL TRIAL: NCT04492579
Title: Neonates Supplemented With Gentle-UHT Donor Human Milk in the First Week of Life
Brief Title: Newborns Supplemented With Gentle-UHT Donor Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LactaLogics, Inc (Industry)
Collaborators: Renown Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5642622173
Record Dates: First submitted 2020-07-23; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Newborns; Breast Milk Expression
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supplementation of Gentle-UHT donor milk (Experimental): Supplementation of Gentle-UHT donor milk in addition to mother's own milk, as recommended by the health care providers.
  Interventions: Other: Gentle-UHT donor human milk supplementation

INTERVENTIONS:
Other: Gentle-UHT donor human milk supplementation — Providers referred mothers with newborns that fit the following criteria: exhibited insufficient milk supply, an infant with early weight loss born >36 weeks gestation. Mother was given Gentle-UHT donor milk for supplementation, in addition to mother's own milk for the first week of the infant's life after hospital discharge.

SUMMARY:
This study evaluates the effects of providing breastfeeding mothers with Gentle-UHT donor human milk (GHM) after discharge to bridge the gap during delayed onset lactation, to support an exclusive human milk diet and continued breastfeeding through the infant's first week of life. The investigators aim to determine the safety of GHM, and if GHM provided to breastfeeding mothers of outpatient babies with early weight loss will ensure babies adequately gain weight according to age-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age >36 weeks
* Exclusively fed human milk
* Age <96 hours (4 days)

Exclusion Criteria:

* Previous admittance to the neonatal intensive care unit
* Supplementation of any formula

Max Age: 4 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2018-08-03 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2020-01-17 (Actual)

PRIMARY OUTCOMES:
Weight gain | 8-9 days of life
  Average weights compared to WHO data

SECONDARY OUTCOMES:
Exclusive human milk diet | 8-9 days of life
  Rates of infants still on an exclusive human milk diet

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Perry, MD, Principal Investigator — Renown Regional Medical Center
Locations (1):
- LactaLogics, Inc., Port Saint Lucie, Florida, United States

IPD SHARING:
Plan to Share IPD: No